CLINICAL TRIAL: NCT04805541
Title: Detection and Classification of Diabetic Retinopathy From Posterior Pole Images With A Deep Learning Model
Status: Completed | Type: Observational
Sponsor: Ural Telekomunikasyon Sanayi Ticaret Anonim Sirketi (Industry)
Collaborators: Akdeniz University (Other)
Responsible Party: Sponsor
Other Study IDs: EC-2021DR-TR
Record Dates: First submitted 2021-03-15; First posted 2021-03-18 (Actual); Results first posted 2024-07-15 (Actual); Last update posted 2024-07-15 (Actual); Status verified 2024-01

CONDITIONS: Diabetic Retinopathy; Diabetic Eye Problems; Diabetic Macular Edema
MeSH Terms: conditions — Diabetic Retinopathy | interventions — Mydriatics

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

INTERVENTIONS:
Procedure: Color Fundus Photography — Subjects will undergo fundus photography before and after administration of mydriatic agent.
Drug: Mydriatic Agent — Subjects will be administered mydriatic medication to dilate their pupils.
  Other Names: Tropicamide drops
Device: EyeCheckup - AI Based DR Screening — Screening for existence of "More than mild" or "Vision-threatening" Diabetic Retinopathy, and/or Diabetic Macular Edema.

SUMMARY:
The duration of diabetes is directly related to eye complications. Diabetic retinopathy affects 80 percent of those who have had diabetes for 20 years or more. At least 90% of new cases can be reduced with proper treatment and monitoring of the eyes. The longer a person has diabetes, the more likely it is to develop diabetic retinopathy. Each year in the United States, diabetic retinopathy accounts for 12% of all new cases of blindness. It is also the leading cause of blindness in people between the ages of 20 and 64. The most important complication of diabetes leading to vision loss is diabetic retinopathy. Depending on this, macular edema, bleeding into the retina and vitreous,neovascular glaucoma can cause blindness.

Diabetic retinopathy (DR) is a leading cause of vision-loss globally. Of an estimated 285 million people with diabetes mellitus worldwide, approximately one third have signs of DR and of these, a further one third of DR is vision-threatening DR, including diabetic macular edema (DME). Diabetic retinopathy is a retinal disease that can often be stopped with early diagnosis, but if neglected, it can lead to severe vision loss, including permanent blindness. Diabetes has high morbidity and there are millions of people who should be screened for diabetic retinopathy (DR). Annual eye screening is recommended for all diabetic patients since vision loss can be prevented if DR is diagnosed in its early stages. Currently, the number of clinical personnel trained for DR screening is less than that needed to screen a growing diabetic population. Therefore, the automatic DR screening system will be able to screen more diabetic patients and diagnose them early.

EyeCheckup is an automated retinal screening device designed automatically analyze color fundus photographs of diabetic patients to identify patients with referable or vision threatening DR. This study is designed to assess the safety and efficacy of EyeCheckup.

The study is a single center study to determine the sensitivity and specificity of EyeCheckup to diabetic retinopathy. EyeCheckup is an automated software device that is designed to analyze ocular fundus digital color photographs taken in frontline primary care settings in order to quickly screen for diabetic retinopathy (DR).

DETAILED DESCRIPTION:
This is a prospective study to assess the safety and efficacy of EyeCheckup in screening for DR.

This study was carried out in a single center at Akdeniz University Faculty of Medicine with primary endpoints to determine the sensitivity and specificity of EyeCheckup to diabetic retinopathy in the primary care setting.

Methods and tools to be used in the study:

* Fundus photography with non-mydriatic camera and classification of diabetic retinopathy with artificial intelligence algorithm,
* Evaluation of seven field dilated fundus images by retina specialists and comparison of results for clinical validation of the system.

Clinical and laboratory tests to be performed:

* Fundus photography with a non-mydriatic camera. In this study, no invasive procedure is applied to the patient, the retinal photograph will be taken with a special digital camera called a fundus camera. In patients whose non-mydriatic image cannot be obtained, tropicamide drops will be instilled to dilate the pupil, and then photographs will be taken.
* Pupil dilation will be achieved by instilling Tropicamide drops in both eyes of the patient, and then 4 quadrant photographs of both eyes will be taken with a mydriatic fundus camera.

After exclusions, this study will enroll up to 900 subjects who are diagnosed with diabetes by the endocrinology polyclinic and meet the eligibility criteria. Participants who meet the eligibility criteria will be recruited after obtaining written informed consent from primary health care providers. Subjects will undergo fundus photography per, Food and Drug Administration (FDA) cleared, ophthalmic cameras (product code: HKI). Images will be taken according to a specific EyeCheckup imaging protocol provided to the ophthalmic camera operator and then analyzed by the EyeCheckup device.

The photography protocol consists of two images of the ocular fundus (one optic disc nerve centered, one macula centered), obtained from both eyes of enrolled participants.

After the retinal images taken from ophthalmic cameras (product code: HKI), images are analyzed with EyeCheckup and a scan report is prepared. If it is necessary to enlarge the pupils, eye enlarging eye drops are applied and wait 15-30 minutes. This information is noted. DR is diagnosed by examination by a retina specialist with the captured images. EyeCheckup success rate is calculated by comparing both reports.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of diabetes mellitus
* Understanding of study and provision of written informed consent
* 18 years of age or older
* No history of any other retinal vascular disease, glaucoma, or other disease that may affect the appearance of the retina or optic disc (refractive error and ocular surface disease are allowed)
* Other than cataract surgery, no history of intraocular surgery, ocular laser treatments for any retinal disease, or ocular injections for diabetic macular edema or proliferative disease No media opacity precluding good retinal photography

Exclusion Criteria:

* No diagnosis of diabetes mellitus
* Potential subject cannot understand study or informed consent
* A history of retinal vascular disease other than diabetic retinopathy that may affect the appearance of the retina or optic disc
* Previous intraocular surgery including cataract; previous laser to the retina; or previous intraocular injections for the treatment of diabetic retinopathy
* Pregnant women or women with gestational diabetes mellitus
* A media opacity in either eye that is severe enough to preclude good retinal photography
* Permanent vision impairment in one or both eyes
* The participant is contraindicated for imaging with fundus imaging systems used in the study:
* Participant is hypersensitive to light
* Participant recently received photodynamic therapy (PDT)
* Participant uses drugs that cause photosensitivity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * Primary care clinic - invitation to volunteer,
  * Diabetic Patients
  * Eighteen years of age or older
  * Have been referred to an ophthalmologist for eye examination to screen for diabetic retinopathy
  * Diseases Polyclinic with the diagnosis of diabetes and were able to view the posterior polar region of the eye with an ophthalmic camera.
    900 volunteer patients who applied to the Akdeniz University Endocrinology and Metabolic
Sampling Method: Non-Probability Sample
Enrollment: 900 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-07-04 (Actual); Study Completion 2022-07-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: A Burak Bilgin, Assoc. Prof., Principal Investigator — Instructor, Retinal Surgeon, Academic Advisor
Locations (1):
- Akdeniz University Hospital, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
No individual data will be shared.

REFERENCES:
- [Derived] Aydemir M, Bilgin AB, Sari R, Dogan ME, Bulut M, Akar Y. Assessment of Correlation Between Diabetic Retinopathy and Metabolic Biomarkers Using Artificial Intelligence. J Diabetes Res. 2026 Jan 14;2026:9085827. doi: 10.1155/jdr/9085827. eCollection 2026. PMID 41541002
- [Derived] Dogan ME, Bilgin AB, Sari R, Bulut M, Akar Y, Aydemir M. Head to head comparison of diagnostic performance of three non-mydriatic cameras for diabetic retinopathy screening with artificial intelligence. Eye (Lond). 2024 Jun;38(9):1694-1701. doi: 10.1038/s41433-024-03000-9. Epub 2024 Mar 11. PMID 38467864

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were reffered to by the Endocrionlogy Department at Akdeniz University Hosptital for an ophthalmic examitation to the opthalmology department to screen for diabetic retinopathy, where they were invited to participate in the study.
Pre-assignment Details: Participants were evaluated for media opacity and other retinal diseases that might prevent good retinal photography.
Groups:
- Screening Population: Prospective Study Participants
Period: Overall Study
Arm/Group | Screening Population
Started | 900
Completed | 865
Not Completed | 35
Not completed — Unable to be retinally photographed with good quality. | 35

BASELINE CHARACTERISTICS:
Population: Number of Enrolled Adult Diabetic Participants
Arm/Group | Screening Population
Number analyzed (Participants) | 900
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.33 (11.16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Sex: Female | 442
  Sex: Male | 458
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Turkey | 900

OUTCOME MEASURES:

1. Primary Outcome: Sensitivity(mtmDR)
Description: Sensitivity for detecting more than mild diabetic retinopathy
Time Frame: 1 visit (1 day)
Measure: Number (95% Confidence Interval); unit: percentage of true positives
Groups:
- Prospective Study Participants (Optomed): Participants Photographed Using Optomed Aurora
- Prospective Study Participants (Canon): Participants Photographed Using Canon CR2
- Prospective Study Participants (Topcon): Participants Photographed Using Topcon NW400
Arm/Group | Prospective Study Participants (Optomed) | Prospective Study Participants (Canon) | Prospective Study Participants (Topcon)
Number analyzed (Participants) | 865 | 704 | 585
percentage of true positives | 90.48 [83.95 to 94.98] | 95.65 [90.15 to 98.57] | 95.19 [89.13 to 98.42]

2. Primary Outcome: Sensitivity(vtDR)
Description: Sensitivity for detecting vision threatening diabetic retinopathy
Time Frame: 1 visit (1 day)
Measure: Number (95% Confidence Interval); unit: percentage of true positives
Arm/Group | Prospective Study Participants (Optomed) | Prospective Study Participants (Canon) | Prospective Study Participants (Topcon)
Number analyzed (Participants) | 865 | 704 | 585
percentage of true positives | 95.12 [87.98 to 98.65] | 96.00 [88.75 to 99.17] | 96.34 [94.56 to 97.67]

3. Primary Outcome: Specificity(mtmDR)
Description: Specificity for detecting more than mild diabetic retinopathy
Time Frame: 1 visit (1 day)
Measure: Number (95% Confidence Interval); unit: percentage of true negatives
Arm/Group | Prospective Study Participants (Optomed) | Prospective Study Participants (Canon) | Prospective Study Participants (Topcon)
Number analyzed (Participants) | 865 | 704 | 585
percentage of true negatives | 97.21 [95.73 to 98.29] | 95.92 [93.99 to 97.37] | 95.93 [93.85 to 97.47]

4. Primary Outcome: Specificity(vtDR)
Description: Specificity for detecting vision threatening diabetic retinopathy
Time Frame: 1 visit (1 day)
Measure: Number (95% Confidence Interval); unit: percentage of true negatives
Arm/Group | Prospective Study Participants (Optomed) | Prospective Study Participants (Canon) | Prospective Study Participants (Topcon)
Number analyzed (Participants) | 865 | 704 | 585
percentage of true negatives | 98.82 [97.77 to 99.45] | 96.34 [94.56 to 97.67] | 95.93 [93.86 to 97.47]

5. Secondary Outcome: Diagnosability
Description: percentage of patients with image quality sufficient for EyeCheckup to produce an output to patients with image quality sufficient for the clinical reference standard to produce an output
Time Frame: 1 Day
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Prospective Study Participants (Optomed) | Prospective Study Participants (Canon) | Prospective Study Participants (Topcon)
Number analyzed (Participants) | 865 | 704 | 585
percentage of participants | 96.57 [96.45 to 98.58] | 100 [99.47 to 100] | 100 [99.37 to 100]

6. Secondary Outcome: Non-Dilated EyeCheckup Usage
Description: Percentage of participants for whom Non-Dilated Images were sufficient to use EyeCheckup
Time Frame: 1 Day
Measure: Number (95% Confidence Interval); unit: percentage of patients imaged undilated
Arm/Group | Prospective Study Participants (Optomed) | Prospective Study Participants (Canon) | Prospective Study Participants (Topcon)
Number analyzed (Participants) | 865 | 704 | 585
percentage of patients imaged undilated | 62.24 [58.88 to 65.52] | 68.90 [65.32 to 72.29] | 78.46 [74.90 to 81.72]

ADVERSE EVENTS:
Time Frame: patient was seen only once for a signle day for retinal imaging throughout the study, therefore 1 day
Description: The images used in our study do not pose any risk or harm to the patients.Only fundus images of the patients will be evaluated.
  The study is expected to pose minimal risk to both camera operators and participants, as the camera systems used have been previously approved by the FDA for ocular fundus photography, and tropicamide 1% eye drops for pupil dilation is an FDA-approved drug product and have been shown to have minimal side effects.
Groups:
- Prospective Study Participants: Screening Population at Primary Care
Arm/Group | Prospective Study Participants
All-Cause Mortality (participants affected / at risk) | 0/865
Serious Adverse Events (participants affected / at risk) | 0/865
Other Adverse Events (participants affected / at risk) | 0/865

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-10-05): https://cdn.clinicaltrials.gov/large-docs/41/NCT04805541/Prot_SAP_000.pdf